CLINICAL TRIAL: NCT03824873
Title: Internal Iliac Artery Ligation Before Cesarean Hysterectomy in Morbidly Adherent Placenta: A Randomized Clinical Trial
Brief Title: Internal Iliac Artery Ligation Before Cesarean Hysterectomy in Morbidly Adherent Placenta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AS1862
Record Dates: First submitted 2019-01-26; First posted 2019-01-31 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Blood Loss
Keywords: Internal iliac artery; Internal iliac artery ligation; Placenta previa; Placenta accreta; cesarean hysterectomy
MeSH Terms: conditions — Hemorrhage; Placenta Previa; Placenta Accreta

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal iliac artery ligation + cesarean hysterectomy (Active Comparator)
  Interventions: Procedure: Internal iliac artery ligation; Procedure: cesarean hysterectomy
- cesarean hysterectomy (Active Comparator)
  Interventions: Procedure: cesarean hysterectomy

INTERVENTIONS:
Procedure: Internal iliac artery ligation — Internal iliac artery ligation and cesarean hysterectomy
  Other Names: cesarean hysterectomy
  Arms: internal iliac artery ligation + cesarean hysterectomy
Procedure: cesarean hysterectomy — cesarean hysterectomy

SUMMARY:
40 pregnant females at term diagnosed with morbidly adherent placenta and planned for elective cesarean section were recruited and randomized to 2 groups. Group A: Internal iliac ligation followed by cesarean hysterectomy. Group B: cesarean hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Placenta previa accreta
* Previous 2 cesarean section
* completed her family
* Hemoglobin > 11 gm/dl
* Elective cesarean hysterectomy

Exclusion Criteria:

* Anemia ( Hemoglobin < 11 gm/dl)
* Not completed her family
* BMI > 35 Kg/m2
* Bleeding tendency
* Emergengy cesarean section
* Thrombophilia

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Amount of blood loss | intraoperative
Amount of Blood transfusion needed in mililiters | 24 hours

SECONDARY OUTCOMES:
change of hemoglobin | 24 hours
change of hematocrit | 24 hours
operative time | intraoperative
incidence of injury of important structures during operation | intraoperative
  incidence of injury of important structures during operation as urinary bladder, ureteric, intestinal or great vessels injury

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No